CLINICAL TRIAL: NCT05041920
Title: A Single-centre, Single-arm, Open-label and Fixed-sequence Study to Evaluate the Effect of Omeprazole on Pharmacokinetics of Famitinib Malate in Healthy Adult Subjects
Brief Title: A Drug-drug Interaction Study of Famitinib Malate With a Proton Pump Inhibitor in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FMTN-I-111
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single-arm, open-label and fixed-sequence drug interaction study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): The study will have only one study group in a fixed-sequence type of design.
  Interventions: Drug: famitinib、omeprazole

INTERVENTIONS:
Drug: famitinib、omeprazole — famitinib malate, 25 mg on study day 1; omeprazole, 40 mg, qd on study day 10-14, 16-22; famotine malate together with omeprazole, on study day 15.

SUMMARY:
The primary objective is to evaluate the effect of omeprazole on the pharmacokinetics of famitinib malate in healthy adult subjects.

The secondary objective is to evaluate the safety after famitinib malate alone or combined administration with omeprazole in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Participants should sign the informed consent before the study, and fully understand the content, process and possible adverse reactions of the study;
2. Capable to complete the study according to the requirements of study protocol;
3. Healthy male and female subjects aged between 18 and 45 (inclusive) at the time of signing the informed consent, of which no less than 1/3 are female subjects;
4. Participants should have no fertility plan from signing the informed consent until 6 months after the last medication, take effective contraceptive measures voluntarily and have no sperm donation plan. The serum HCG test of fertile women must be negative before Screening;
5. Body weight ≥ 50.0 kg for men and body weight ≥ 45.0 kg for women, and body mass index (BMI) within the range of 19.0 to 28.0 kg /m2 (inclusive);
6. Creatinine clearance (CLCr) ≥80 mL/min, and creatinine is less than or equal to the upper limit of normal value.

Exclusion Criteria:

1. Those who donated blood or suffered blood loss ≥400 mL within 3 months prior to Screening, donated blood or suffered blood loss ≥200 mL within 1 month prior to Screening, or received blood transfusion;
2. Allergic constitution, including a history of severe drug/food allergy; Any history of allergy to famitinib malate capsules or omeprazole magnesium enteric-coated tablets;
3. Any history of drug abuse, positive results for alcohol, nicotine or drugs at Screening;
4. Those who have heavy smokers and alcoholic will not be able to prohibit smoking and alcohol during the trial;
5. Any history of dysphagia or any gastrointestinal disease that affects drug absorption;
6. Those who have any uncontrolled peptic ulcer, colitis, pancreatitis, etc.;
7. Those who have received any operation within 6 months before Screening; Previous surgery affecting gastrointestinal absorption (including gastrectomy, intestinal resection, gastric contraction surgery, etc.);
8. Subjects with any clinically significant acute disease occurring within 1 month prior to Screening;
9. QTcF>470 msec for women or >450 msec for men;
10. Any pre-existing chronic or severe medical history of nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolism, and musculoskeletal system;
11. Participation in any clinical trial within 3 months before Screening;
12. Those who took any other drugs that affect liver metabolism within 28 days prior to taking the investigational drug;
13. Those who took any prescription or non-prescription drugs, any vitamin products or herbal medicine within 14 days prior to receiving the investigational drug;
14. Abnormal vital signs at Screening;
15. Clinical laboratory tests, infectious disease screening, 12-lead electrocardiogram, abdominal B ultrasound, X-ray or CT examination with abnormalities and clinical significance;
16. Consumption of grapefruit or grapefruit products, caffeine, or xanthine foods or beverages within 48 hours prior to taking the investigational drug; Strenuous exercise, or other factors affecting drug absorption, distribution, metabolism, excretion, etc.;
17. Lactating women;
18. History of injection needle or blood fainting, those who have difficulty in blood collection or cannot tolerate venepuncture blood collection; Those who cannot accept a uniform diet;
19. Subjects with other factors unsuitable to participate in the study considered by the researcher or subjects withdraw from the study due to their own reasons.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Cmax | day 1 to day 23
AUC0-t | day 1 to day 23
AUC0-∞(if applicable) | day 1 to day 23
Tmax | day 1 to day 23
t1/2 | day 1 to day 23
CL/F | day 1 to day 23
Vz/F | day 1 to day 23

SECONDARY OUTCOMES:
The incidence and severity of adverse events/serious adverse events | from ICF signing date to approximate day 30

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, Affiliated to Southest University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided